CLINICAL TRIAL: NCT02213835
Title: Treatment With the Specific Carbohydrate Diet for Children With Active Crohns Disease and Ulcerative Colitis
Acronym: SCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Suskind (Other)
Responsible Party: Sponsor-Investigator, David Suskind, Professor of Pediatrics, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCD001
Record Dates: First submitted 2014-08-04; First posted 2014-08-12 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2018-05

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Crohn's disease and Ulcerative colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Specific Carbohydrate diet (SCD) (Experimental): The treatment for this study will be the Specific Carbohydrate diet (SCD). Intervention will be based upon standard dietary therapy as well as a nutritional handbook developed in the Gastroenterology division. Patients will receive one-on-one guidance by a Seattle Children's Dietician trained in the SCD during each visit. Prior to each visit patient will fill out a 3 day nutrition log which will be reviewed by the dietician during the clinic visit. Each patient will receive books on the SCD therapy which will include recipes and information about the diet The two books given will include "Breaking the Vicious Cycle" by Elaine Gottschall and "Recipes for the Specific Carbohydrate Diet" by Raman Prasad.
  Interventions: Other: Specific Carbohydrate diet (SCD)

INTERVENTIONS:
Other: Specific Carbohydrate diet (SCD)

SUMMARY:
The aim of this study is to determine the tolerability and potential efficacy of dietary therapy, the Specific Carbohydrate Diet (SCD), in pediatric patients with Crohn's disease (CD) and Ulcerative Colitis (UC). This is a single center, open labelled study designed to determine tolerability, preliminary safety and potential efficacy in pediatric patients with CD and UC. The study patients will be recruited from Seattle Children's GI clinic. the investigators will enroll 10 patients with mild to moderate CD (defined as PCDAI score of 10-29) or Ulcerative colitis (PUCAI 10-60) ages 8 to 21 years. Each patient will be in the study for approximately 12 weeks.

DETAILED DESCRIPTION:
Ten patients with CD or UC with mild or moderate disease activity as defined by Pediatric Crohn's disease activity index (PCDAI score of 10-29 or PUCAI of 10 - 60) aged 8 -21 years will enroll into this study. Each patient will receive an initial evaluation including a physical exam, medication review, nutritional guidance and post treatment evaluations.

Initial evaluation: Study subject recipient will have the following lab tests including CBC with differential & platelets, a c-reactive protein, sedimentation rate, an albumin, vitamin D level, a stool study for c. difficile, for bacterial culture and ova and parasite, stool calprotectin and microbiome. Additionally, the investigators will complete a physical exam and document their current medications. The study nutritionist will complete a thorough diet history.

Treatment: The treatment for this study will be the Specific Carbohydrate diet (SCD). Intervention will be based upon standard dietary therapy as well as a nutritional handbook developed in the Gastroenterology division. Patients will receive one-on-one guidance by a Seattle Children's Dietician trained in the SCD during each visit. Prior to each visit patient will fill out a 3 day nutrition log which will be reviewed by the dietician during the clinic visit. Each patient will receive books on the SCD therapy which will include recipes and information about the diet The two books given will include "Breaking the Vicious Cycle" by Elaine Gottschall and "Recipes for the Specific Carbohydrate Diet" by Raman Prasad.

Follow-up: Each study subject will have clinical follow-up at 2 weeks, 4 weeks, 8 weeks and 12weeks. Standardized questionnaires, including the Pediatric Crohn's disease activity index (PCDAI) or Pediatric Ulcerative colitis activity index (PUCAI) will be completed during each study visit. Information about tabulating the PCDAI/PUCAI scores is listed in Appendix A. In addition patients will have a physical exam and standard blood work including CBC, sedimentation rate, C-reactive protein, albumin and stool for microbiome analysis at each follow up visit. This stool will be sent to the University of Washington (Dr. Sam Miller's lab) for analysis. Stool calprotectin will additionally be done at week 4 and 12. Vitamin D level will be measured at week 12. Finally, all patients will meet with the nutritionist at each visit who will complete a thorough diet review. Any questions about the SCD will be addressed at each visit.

All study related information will be stored in the RedCap database. Participant data for the study will be stored electronically in the REDCap platform. The REDCap platform is managed by the Institute for Clinical and Translational Science at the University of Washington. Only IRB approved research team members will have access to the REDCap data platform. Each team member will be granted access to the REDCap data system through a secure login. The information about each participant will be de-identified using a unique study code. Some personal information such as date of birth will be stored in RedCap.

Microbiome:

Some stool from the participants at screening, week 2, 4, 8 and 12 will be stored for microbiome analysis. The samples will be stored at Seattle Children's Hospital in the Clinical Research Center lab in the -80 freezer. These samples will be sent to the University of Washington for microbiome analysis and storage on an as necessary basis. Each of these samples will be de-identified and labeled with a unique study code and visit number. Consent for storage will be part of the Informed Consent process.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescents eight to twenty one years old
2. Diagnosis of Ulcerative colitis or Crohn's Disease made by a primary gastroenterologist based upon history, physical exam, laboratory/radiological studies and gastrointestinal histology
3. Mild or moderate disease activity based upon PCDAI score (10-45) or PUCAI score (10-60)
4. Parent/guardian and child must be able to comprehend the consent and assent
5. Parent/guardian and participant must be able to attend study visits at baseline, and weeks +2, +4, +8, +12.
6. Patient must not have medication changes for his/her inflammatory bowel disease medications for at least 1 months, unless medically necessary.

Exclusion Criteria:

1. Severe disease with PCDAI >45 or PUCAI >60
2. Active or history of intraabdominal abscess, intraabdominal fistula, stricturing Crohn's disease
3. Other serious medical conditions such as neurological, liver, kidney, autoimmune or systemic disease.
4. Has begun TNF inhibitors within two months prior to study
5. Has had change of maintenance medication within the last month
6. Tobacco, alcohol or illicit drug abuse
7. Pregnant subject recipients will be excluded

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2014-06; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in Pediatric Crohn's disease Activity Index/Pediatric Ulcerative Colitis Activity Index at baseline and 12 weeks | 12 Week
  Pediatric Crohn's disease Activity Index/Pediatric Ulcerative Colitis Activity Index are validated measures of disease activity for pediatric Crohn's disease and ulcerative colitis respectively.

SECONDARY OUTCOMES:
Change of common Laboratory measures including Complete Blood Count, sedimentation rate, C-Reactive Protein, stool Calprotectin at baseline and 12 weeks | 12 weeks
  Validated clinical laboratory tests preformed at an accredited laboratory

OTHER OUTCOMES:
Stool Microbiome Analysis from baseline and 12 weeks | 12 Weeks
  Changes in fecal microbiome as defined by species types and percent of total microbiome will be measured using Metagenomic Phylogenetic Analysis (MetaPhlAn)

CONTACTS AND LOCATIONS:
Overall Officials: David L Suskind, MD, Principal Investigator — Seattle Children's Hospital and The University of Washington
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Not discussed

REFERENCES:
- [Background] Suskind DL, Wahbeh G, Gregory N, Vendettuoli H, Christie D. Nutritional therapy in pediatric Crohn disease: the specific carbohydrate diet. J Pediatr Gastroenterol Nutr. 2014 Jan;58(1):87-91. doi: 10.1097/MPG.0000000000000103. PMID 24048168
- [Derived] Braly K, Williamson N, Shaffer ML, Lee D, Wahbeh G, Klein J, Giefer M, Suskind DL. Nutritional Adequacy of the Specific Carbohydrate Diet in Pediatric Inflammatory Bowel Disease. J Pediatr Gastroenterol Nutr. 2017 Nov;65(5):533-538. doi: 10.1097/MPG.0000000000001613. PMID 28825603